CLINICAL TRIAL: NCT02863549
Title: Transcatheter Treatment of Severe Tricuspid Regurgitation Using the MitraClip System
Brief Title: MitraClip for Severe TR
Acronym: TVrepair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Daniel Braun, MD, MD, Attending Physician, LMU Klinikum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MucS001-17
Record Dates: First submitted 2016-07-20; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MitraClip in tricuspid valve — MitraClip in tricuspid valve

SUMMARY:
The aim of this study was to investigate the procedural feasibility and 30-day results of transcatheter tricuspid valve repair using the MitraClip® system (Abbott Vascular) in selected, highly symptomatic patients with severe tricuspid regurgitation (TR).

DETAILED DESCRIPTION:
The primary objectives of this prospective analysis were to determine the feasibility in terms of success rate and short-term clinical follow-up at 30 days. In this context procedural success was defined as reduction of at least one TR grade. At 30-days after the procedure, a clinical follow up was performed in the heart failure outpatient clinic of our department including transthoracic echocardiography for the evaluation of TR grades. Furthermore, the investigators determined NYHA functional class and the incidence of major adverse cardiac and cerebrovascular events (MACCE).

Secondary objectives were the assessment of right ventricular function, the 6-minute walk distance, NT-proBNP as well as quality of life as assessed by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) score at 30-days follow up.

ELIGIBILITY:
Inclusion Criteria:

* right-sided heart failure due to moderate-to-severe tricuspid regurgitation
* patients deemed inoperable by the heart Team

Exclusion Criteria:

* poor Echo-image quality

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
TR grade, Echo (grade 0-4) | 1-12 months
  grade 0-4: 0: no tricuspid regurgitation, 4: massive TR
MACCE | 1-12 months

SECONDARY OUTCOMES:
NYHA status | 1-12 months
6 Minute walk distance | 1-12 months
NT-proBNP | 1-12 months
MLHFQ | 1-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Braun, MD, Principal Investigator — Klinikum der Universität München
Locations (1):
- Klinikum Großhadern University Hospital, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No